CLINICAL TRIAL: NCT00501345
Title: Effects of Aspirin on Platelet Function and Clinical Outcome in Patients With Thrombocytopenia, Neoplasm, and Myocardial Infarction
Brief Title: Aspirin in Patients With Myocardial Infarction and Thrombocytopenia
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Low accrual, study terminated.
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ID01-674
Record Dates: First submitted 2007-07-13; First posted 2007-07-16 (Estimated); Results first posted 2010-10-13 (Estimated); Last update posted 2012-08-01 (Estimated); Status verified 2012-07

CONDITIONS: Thrombocytopenia; Myocardial Infarction
Keywords: Thrombocytopenia; Platelet Function; Acute Coronary Syndrome; Myocardial Infarction; Heart Attack; Aspirin
MeSH Terms: conditions — Thrombocytopenia; Myocardial Infarction; Acute Coronary Syndrome | interventions — Aspirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Aspirin (Experimental)
  Interventions: Drug: Aspirin

INTERVENTIONS:
Drug: Aspirin — 325 mg by mouth on Day 1 only, followed by 160 mg by mouth daily

SUMMARY:
Primary Objective:

To determine the risk of bleeding from ASA therapy in thrombocytopenic patients who develop Acute Coronary Syndrome (ACS), and assess its effect on the overall morbidity and mortality in these patients as well as platelet functions.

DETAILED DESCRIPTION:
Aspirin is known to decrease death rate by as much as 50% in patients that suffer from heart attacks. Patients with low platelet count are not given aspirin for fear of an increased risk of bleeding. Researchers want to compare the risks versus the benefits of using aspirin in this patient population.

Participants in this study who suffer chest pain will be treated with a single enteric coated aspirin 325 mg instead of the current treatment without aspirin. Participants will then be tested to confirm that they had a heart attack by EKG (a test to measure the electrical activity of the heart) and blood tests (5ml of blood) will be drawn every 8 hours to detect enzymes that are released from the heart due to the heart attack. Blood samples will also be examined for platelet number.

Participants who are found to have had a heart attack and have a platelet count of between 100,000 and 20,000 will be continued on aspirin (160 mg per day). All other standard medications for heart attacks will also be given.

Participants who are found to have had a heart attack but whose platelet number is more than 100,000 will be given the standard therapy for heart attack, including enteric coated aspirin 325 mg per day, and will no longer take part in this study. Participants who are found to have had a heart attack but whose platelet number is less than 20,000 will be not be included in the study and will be treated as deemed appropriate by their primary physician.

Participants will be examined daily and evaluated for bleeding. Blood samples (30 ml of blood) will also be drawn before or after aspirin is given and 24 hours, 72 hours and 7 days after aspirin treatment to study platelet function. Participants will be followed up on the study for 7 days. Participants will be followed up in the cardiology clinic within 1-2 weeks after discharge from the hospital, then once a month for six month. Further follow up will be every 6 month. Patients are requested to follow up with cardiology by phone at any time for any bleeding.

Participants who are not found to have had a heart attack will not receive any further aspirin treatment.

This is an investigational study. Aspirin is an FDA approved drug for treatment of heart attacks and is commercially available. Aspirin is a standard therapy for patients who have had a heart attack. Thirty patients will take part in this study. All will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Presenting for Cardiology consult at M.D. Anderson Cancer Center.
2. Platelet count between 100,000 and 20,000.
3. Acute Coronary Syndrome diagnosed with their first 12 lead EKG.
4. Patients that continue to show evidence of MI by cardiac enzymes with CPK levels > 2 normal limits, CK-MB levels 10% above normal limits, and Troponin I levels > 1.4ug/L will be considered positive for MI.
5. Ability to give consent.

Exclusion Criteria:

1. Contraindications to aspirin including severe intolerance or true allergy, active bleeding, hemophilia, active retinal bleeding, severe untreated hypertension, active peptic ulcer, or other significant source of gastrointestinal or genitourinary bleeding, brain metastasis, and altered mental status.
2. Unwillingness or inability to give consent.
3. Progressive heart failure, unstable angina not responding to medical therapy for 24 hours, or ventricular tachycardia, necessitating thrombolysis, and angioplasty.
4. Patients that rule out for MI by cardiac enzymes panel after the first 24 hours.
5. Patients that rule in for MI and have Platelet count > 100,000.
6. Patients with platelet count < 20,000.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2002-02; Primary Completion 2008-02 (Actual); Study Completion 2008-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Bernard Durand, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- U.T.M.D. Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: The University of Texas M.D.Anderson Cancer Center — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: 02/28/02 through 04/22/04. All participants recruited at UT MD Anderson Cancer Center.
Pre-assignment Details: Study terminated as a result of difficulty in accrual of candidate patients for enrollment. Six patients were enrolled but one patient did not meet eligibility criteria.
Groups:
- Aspirin: 325 mg by mouth Day 1, 160 mg daily thereafter
Period: Overall Study
Arm/Group | Aspirin
Started | 5
Completed | 5
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Aspirin
Number analyzed (Participants) | 5
Age Continuous [Median (Full Range); unit: years] | 78 [39 to 88]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 3
Region of Enrollment [Number; unit: participants]
  United States | 5

OUTCOME MEASURES:

1. Primary Outcome: Participants With 7 Days Observation Without Severe Bleeding
Description: Blood samples collected at baseline before or after aspirin is given and at 24 hours, 72 hours and 7 days after treatment has been initiated for those that remain in the study after the first 24 hours.
Time Frame: 7 Days
Population: The baseline Thromboelastogram showed normal platelet function in all patients and no evidence of heparin induced thrombocytopenia (HIT). No further analysis was done as study was terminated due to lack of accrual.
Arm/Group | Aspirin
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 2 Years
Arm/Group | Aspirin
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

LIMITATIONS AND CAVEATS:
A change in hospital practice where patients with thrombocytopenia now routinely receive aspirin for acute coronary syndromes makes it difficult to obtain a baseline thromboelastogram.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No